CLINICAL TRIAL: NCT06254508
Title: The Effectiveness of an Online FITT-VP Principle Based Exercise Program and Dietary Guidance in the Management of Childhood and Adolescent Obesity.
Brief Title: Online Exercise Program and Dietary Advice (FITT-online) for Children and Adolescents With Obesity
Acronym: FITT-online
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Shanghai Simlab Health Technology (Unknown)
Responsible Party: Principal Investigator, Feihong Luo, Chief, Department of Endocrinology and Inherited Metabolic Diseases, Children's Hospital of Fudan University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FITT-online-[2023]-251
Record Dates: First submitted 2024-01-26; First posted 2024-02-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FITT to CON (Active Comparator): Online program that includes exercise guided by the FITT-VP principle and dietary advice for 16 weeks, followed by conventional in-clinic nutrition and exercise advice and self-control for 16 weeks.
  Interventions: Behavioral: Online program that includes exercise guided by the FITT-VP principle and dietary advice; Behavioral: Conventional in-clinic nutrition and exercise advice and self-control
- CON to FITT (Active Comparator): Conventional in-clinic nutrition and exercise advice and self-control for 16 weeks, followed by online program that includes exercise guided by the FITT-VP principle and dietary advice for 16 weeks.
  Interventions: Behavioral: Online program that includes exercise guided by the FITT-VP principle and dietary advice; Behavioral: Conventional in-clinic nutrition and exercise advice and self-control

INTERVENTIONS:
Behavioral: Online program that includes exercise guided by the FITT-VP principle and dietary advice — 1. Week 1: Children received 2 sessions of exercise initiation and 1 session of small group exercise training (45 minutes) with 4~6 peers.
  2. Weeks 2 to 16: 3 small group exercise sessions per week (45 minutes, 4-6 peers) of moderate-to-vigorous physical activity (MVPA). Effective exercise time was assessed by the time subjects reached the heart rate corresponding to the exercise intensity (64-95% of maximal heart rate), as measured by the instantaneous heart rate recorded during each exercise session. The type of exercise was a combination of aerobic, resistance, and flexibility exercises (time ratio 2.5:1:1).
  3. Dietary guidance was provided concurrently during the 16-week intervention period: by establishing a WeChat group for caregivers and uploading daily pictures of the day's food to the group, the group's health coaches provided daily targeted dietary guidance.
Behavioral: Conventional in-clinic nutrition and exercise advice and self-control — Physicians provide instructions on exercise and nutrition (total daily calorie intake) for the patients to conduct self-control for 16 weeks.

SUMMARY:
This controlled clinical trial aims to compare the effects of an online program that includes exercise guided by the FITT-VP principle and dietary advice, conducted by fitness coaches, in children and adolescents with obesity with a control group that will be enrolled in conventional in-clinic nutrition and exercise advice. All participants will be monitored for 8 months during the active intervention, and followed by 16 months of observation.

The study will evaluate the following parameters between groups: BMI, anthropometry, blood biochemistry panel (ALT/AST, lipids, uric acid, HOMA-IR, HbA1c), food frequency questionaire, household survey, satisfaction survey, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Simple obesity: Body mass index (BMI) between +2SD and +3SD of the reference range: based on the "Standard Deviation Curve of BMI for Children 0-18 Years of Age in China", which was developed by the Physical Development Survey of Children in Nine Provinces/Cities in 2005;
2. Not participating in other weight management programs currently or in the 3 months prior to the study;
3. Accepts to participate and signs informed consent.

Exclusion Criteria:

1. Currently taking or planning to take medications or interventions that affect body weight during the study period (32 weeks)
2. Obesity caused by other medical conditions. For example, hypothalamic-pituitary disease, hypothyroidism, growth hormone deficiency, Cushing's syndrome, obesity-related syndromes.
3. Comorbidity with other chronic diseases. E.g. psychiatric diseases, respiratory diseases, gastrointestinal diseases, rheumatic diseases, hepatic and renal insufficiency, chronic infectious diseases;
4. Presence of abnormal laboratory values at the time of screening indicating a clinically significant underlying disease or condition that may prevent the subject from participating in the study; or presence of abnormalities in the following laboratory tests: alanine aminotransferase (ALT) greater than 5 times the upper limit of normal, serum creatinine (Scr) greater than 1.5 times the upper limit of normal.
5. Contraindications to physical exercise or exercise-related risks. For example, history of asthma, history of hypoglycemia/diabetes, history of heart disease, history of cardiovascular disease, fracture/surgery/planned surgery within the last 1 year, psychomotor retardation, motor system defects/disabilities, previous history of exercise intolerance;

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
BMI | 16, 32, 52, 104 weeks
  Reduction in body mass index (the body mass [kg] divided by the square of the body height [m])

SECONDARY OUTCOMES:
Dietary habits | 16, 32, 52, 104 weeks
  Change in dietary habits assessed by food frequency questionaire (2015 CHNS)
AE | 16, 32, 52, 104 weeks
  Adverse events during active intervention by questionaire and healthcare records according to local regulations (PMID: 34327433)
Uric acid | 16, 32 weeks
  Reduction in serum uric acid levels
Tch | 16, 32 weeks
  Reduction in serum total cholesterol
LDL-c | 16, 32 weeks
  Reduction in serum low density lipoprotein cholesterol
HbA1c | 16, 32 weeks
  Reduction in glycated hemoglobin
HOMA-IR | 16, 32 weeks
  Reduction in this surrogate marker of beta-cell function and insulin resistance (IR) from basal (fasting) glucose and concentrations.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No